CLINICAL TRIAL: NCT04729582
Title: Combined Phase 1 and 1/2a Clinical Trial Evaluating the Safety and Efficacy of an Autologous Muscle Stem Cell Therapy in the Treatment of Urinary Incontinence in Isolated Epispadias
Brief Title: Autologous Muscle Stem Cell Therapy for Treatment of Congenital Urinary Incontinence in Epispadias Patients
Acronym: MUST
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Simone Spuler, MD (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Simone Spuler, MD, Principal investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUST
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence; Epispadias, Male
Keywords: Isolated epispadias; Urinary incontinence; Muscle stem cell therapy; Autologous cell therapy
MeSH Terms: conditions — Urinary Incontinence; Epispadias

STUDY DESIGN:
Intervention Model Description: This is a randomized placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Group (Experimental): Participants receive primary human muscle stem cells as one-time injection into the urethral sphincter region under visual control using cystoscopy.
  Interventions: Biological: Primary human muscle stem cells (Satori-01)
- Placebo group (Placebo Comparator): Participants receive placebo solution as one-time injection into the external urethral sphincter region under visual control using cystoscopy.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Primary human muscle stem cells (Satori-01) — Primary human muscle stem cells are isolated from patient's muscle tissue and expanded ex-vivo. They are injected into the urethral sphincter region as a one-time autologous treatment.
  Arms: Verum Group
Other: Placebo — Placebo is the injection solution without muscle stem cells.
  Arms: Placebo group

SUMMARY:
The aim of this trial is to evaluate the safety and efficacy of an autologous muscle stem cell therapy in the treatment of congenital urinary incontinence in isolated epispadias.

DETAILED DESCRIPTION:
Epispadias is the mildest form of exstrophy-epispadias complex (EEC); a congenital malformation disorder involving the midline abdominal and genitourinary structures. Patients with epispadias have a defect in the urethral sphincter resulting in urinary incontinence. This trial investigates the injection of autologous primary human muscle stem cells into the urethral sphincter with the aim of repairing the defect and restore the anatomic ability for continence.

Eligible participants will undergo muscle biopsy during a routine cystoscopy. Acquired muscle tissue is used for the isolation and expansion of muscle stem cells ex-vivo. Muscle stem cells are injected into the urethral sphincter under visual control using cystoscopy. Participants are assessed for safety and efficacy for a minimum of 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Isolated epispadias
* Aged ≥ 3 years
* Urinary incontinence as defined according to the International Children´s Continence Society
* Informed consent

Exclusion Criteria:

* Acute or chronic inflammatory local or systemic disease
* Coagulation Disorder
* Previous adverse reaction to anesthesia
* Congenital heart defect, cardiac arrhythmia

Ages: 3 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Intervention-related Adverse Events | Upto 12 months post-intervention
  Characterization of type, incidence, severity, and duration of adverse events
Change in Leak Point Pressure (LPP) | Six months post-intervention
  Change in LPP is calculated from baseline measurement

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ebert, Prof. Dr., Principal Investigator — Pediatric Urology, Department for Urology University of Ulm, Germany
Locations (2):
- Germany (2):
  - Clinic for Pediatric Urology in cooperation with University Hospital Regensburg, St. Hedwig Hospital, Regensburg
  - Pediatric Urology, Department for Urology University of Ulm, Ulm